CLINICAL TRIAL: NCT06731517
Title: Comparison of Ultrasound and CT-Based Anatomical Measurements with Classical Methods for Predicting Size and Optimal Placement Depth of Left-Sided Double-Lumen Endobronchial Tubes in Thoracic Surgery
Brief Title: Comparison of Ultrasound, CT, and Classical Methods for Selecting Sizes and Placement of Left-Sided Double-Lumen Tubes
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: ANKCHBILKENT-ANES-SO-01
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Thoracic Neoplasms
Keywords: double lumen tube; size; depth; malposition; ultrasonography; computed tomography; fiber optic bronchoscopy
MeSH Terms: conditions — Thoracic Neoplasms | interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Classical group: In the classical group, Double Lumen Tube selection was based on gender and height. For males, a 41 F tube was chosen if height >170 cm, and a 39 F tube if height ≤170 cm. For females, a 37 F tube was used if height >160 cm, and a 35 F tube if height ≤160 cm. The depth was determined using the formula: 12 + (patient height/10). The calculated depth was marked on the DLT, and after intubation, the mark was positioned at the level of the upper teeth.
  Interventions: Procedure: intubation
- Ultrasonography group: In the Ultrasonography (USG) group, Double Lumen Tube selection was based on the transverse cricoid cartilage diameter measured preoperatively using ultrasound. A 41 F tube was selected if the cricoid diameter was ≥18 mm, 39 F for 16-17.9 mm, 37 F for 15-15.9 mm, 35 F for 13-14.9 mm, and 32 F for <13 mm (Table 5) (5). To determine placement depth, the distance between the vocal cords and the Louis angle was measured (the Louis angle was used as a guide as it anatomically aligns with the carina). The position of the vocal cords was identified using USG. The measured length was marked starting from the bronchial cuff line, and this mark was positioned at the level of the vocal cords during intubation.
  Interventions: Procedure: intubation
- Computed Tomography: In the Computed Tomography (CT) group, Double Lumen Tube selection was based on CT measurements. Radiologists measured the cricoid diameter and the distance between the carina and the vocal cords. A 41 F tube was selected if the cricoid diameter was ≥18 mm, 39 F for 16-17.9 mm, 37 F for 15-15.9 mm, 35 F for 13-14.9 mm, and 32 F for <13 mm (Table 5) (5). The calculated depth was marked starting from the bronchial cuff line, and this mark was positioned at the level of the vocal cords during intubation.
  Interventions: Procedure: intubation

INTERVENTIONS:
Procedure: intubation — Double-Lumen Tube Intubation

SUMMARY:
Investigators aimed to compare anatomical measurements obtained using ultrasound and computed tomography with classical methods to select the appropriate size of double-lumen tubes more quickly and easily and to determine the optimal depth of placement.

DETAILED DESCRIPTION:
In modern thoracic anesthesia, one-lung ventilation (OLV) is essential for managing surgeries, and double-lumen tubes (DLTs) have been a key advancement. DLTs allow separate lung ventilation, facilitating lung deflation and preventing material transfer to the healthy lung. However, improper DLT placement can compromise these functions, emphasizing the importance of correct sizing and positioning.

Choosing the right DLT size depends heavily on patient-specific factors. Undersized DLTs can cause airway injuries, increased resistance, and displacement, while oversized DLTs are linked to postoperative issues like sore throat and difficult intubation. Despite this, no universal criterion exists for DLT size selection. Traditional methods rely on height and gender, but weak correlations with airway size often lead to improper choices, especially in shorter individuals.

Imaging techniques like chest X-rays, Computed Tomography (CT), and ultrasonography (USG) offer a more precise approach to airway measurements for DLT selection. USG is especially advantageous due to its accessibility, speed, and ease of use in operating rooms and emergencies. To improve the accuracy and ease of DLT size selection and placement, investigators aimed to compare anatomical measurements from USG and CT with traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* Requiring lung isolation in thoracic surgery,
* American Society of Anesthesiologists (ASA) risk score of 1-2-3,
* Patients who are literate and able to provide informed consent

Exclusion Criteria:

* Patients with an ASA score of 4 or higher,
* Criteria for difficult intubation,
* Difficulty in mouth opening, small jaw deformities,
* Abnormal cricoid cartilage appearance,
* A history of laryngeal or neck surgery,
* Preoperative throat pain and hoarseness,
* Tumors and deformities in the main airway

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: "A total of 150 patients aged 18-80 years, requiring lung isolation in thoracic surgery, with an American Society of Anesthesiologists (ASA) risk score of 1-2-3, who were literate and able to provide informed consent, were included in the study."
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
malposition | 10 minutes
  After intubation in all three groups;
  1. The upper teeth level was checked and the cm was recorded. It was checked whether both lungs were equally ventilated with the inspection and auscultation method. First, the tube lumens were clamped on the left side; it was checked whether the right lung was ventilated, then the same procedure was repeated for the right side and noted. Then, both lungs were ventilated with 6-8 ml/kg tidal volume and the airway pressure was recorded. With the help of the clamp, the left side was clamped first, the right lung was ventilated with 4-6 ml/kg tidal volume and the airway pressure was checked. The same procedure was repeated for the other side. It was determined whether there was sufficient isolation according to the difference between the airway pressures and recorded.
  Isolation criteria:
  Satisfactory isolation: If the respiratory sounds are clearly heard on the opposite side when one lung is isolated and the airway pressure on the other side increa
Appropriateness of the Selected DLT Size | 10 minutes
  The selected tube was evaluated to see if it was of appropriate size.
  Appropriate size: If the double-lumen tube tip entered the left main bronchus and no obvious resistance was encountered and there was no airway leakage and isolation was achieved when the bronchial cuff was inflated with 1-3 ml and the tracheal cuff with 2-6 ml of air, it was accepted that the double-lumen tube was selected in an appropriate size.
  Large tube: If the double-lumen tube tip could not enter the left main bronchus or was placed in the left main bronchus, but when the bronchial cuff was inflated with less than 1 ml and the tracheal cuff with less than 2 ml of air, pulmonary isolation was achieved and there was no air leakage, it was accepted that it was a large-sized double-lumen tube.
  Small tube: If the bronchial cuff was inflated with more than 3 ml and the tracheal cuff with more than 6 ml of air, pulmonary isolation was achieved and there was no air leakage, it was accepted that it was a small-size
Appropriateness of Double-Lumen Tube Placement | 10 minutes
  While the patient was in the supine position, the location of the tube was checked with fiber optic bronchoscopy. It was noted whether the tube was in its optimum location. If not, how many cm it should be advanced or retracted for its optimum location.

SECONDARY OUTCOMES:
Subglottic resistance | 10 minutes
  Subglottic resistance was assessed and recorded as none, mild, moderate, or severe based on the level of resistance.
Petechiae | 10 minutes
  It was noted with FOB whether there were petechiae in the trachea, bronchi, or both.
Hoarseness | 24 hours
  Hoarseness was assessed as follows.
  0: No hoarseness
  1. Hoarseness noticed by the patient
  2. Hoarseness noticed by the observer
  3. Aphonia
Throat Pain | 24 hours
  Throat pain was assessed and recorded 24 hours postoperatively.
  Sore throat; evaluated as follows.
  0: No sore throat
  1. Mild pain with swallowing
  2. Constant pain that increases with swallowing
  3. Severe pain that prevents eating and requires analgesia

CONTACTS AND LOCATIONS:
Overall Officials: SUMRU ŞEKERCİ, PROF, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, ÇANKAYA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Wang DX, Wei JQ, Liu H, Hu SP. Recent advances in double-lumen tube malposition in thoracic surgery: A bibliometric analysis and narrative literature review. Front Med (Lausanne). 2022 Dec 14;9:1071254. doi: 10.3389/fmed.2022.1071254. eCollection 2022. PMID 36590949
- [Background] Chang TR, Yuan MK, Pan SF, Chuang CC, So EC. Double-Lumen Endotracheal Tube-Predicting Insertion Depth and Tube Size Based on Patient's Chest X-ray Image Data and 4 Other Body Parameters. Diagnostics (Basel). 2022 Dec 14;12(12):3162. doi: 10.3390/diagnostics12123162. PMID 36553170
- [Background] Woo JH, Cho S, Kim YJ, Kim DY, Choi Y, Lee JW. Depth of double-lumen endobronchial tube: a comparison between real practice and clinical recommendations using height-based formulae. Anesth Pain Med (Seoul). 2023 Jan;18(1):37-45. doi: 10.17085/apm.22214. Epub 2023 Jan 10. PMID 36746900
- [Background] Shiqing L, Wenxu Q, Yuqiang M, Youjing D. Predicting the Size of a Left Double-Lumen Tube for Asian Women Based on the Combination of the Diameters of the Cricoid Ring and Left Main Bronchus: A Randomized, Prospective, Controlled Trial. Anesth Analg. 2020 Mar;130(3):762-768. doi: 10.1213/ANE.0000000000003839. PMID 30286004
- [Background] Brodsky JB, Macario A, Mark JB. Tracheal diameter predicts double-lumen tube size: a method for selecting left double-lumen tubes. Anesth Analg. 1996 Apr;82(4):861-4. doi: 10.1097/00000539-199604000-00032. No abstract available. PMID 8615510
- [Background] Eldawlatly AA. Double lumen tube: Size and insertion depth. Saudi J Anaesth. 2021 Jul-Sep;15(3):280-282. doi: 10.4103/sja.sja_192_21. Epub 2021 Jun 19. PMID 34764835
- [Background] Liu Z, Zhao L, Jia Q, Yang X, Liang SJ, He W. Chest Computed Tomography Image for Accurately Predicting the Optimal Insertion Depth of Left-Sided Double-Lumen Tube. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):855-859. doi: 10.1053/j.jvca.2017.09.025. Epub 2017 Sep 20. PMID 29221981
- [Background] Zhang C, Qin X, Zhou W, He S, Liu A, Zhang Y, Dai Z, Yin J. Prediction of Left Double-Lumen Tube Size by Measurement of Cricoid Cartilage Transverse Diameter by Ultrasound and CT Multi-Planar Reconstruction. Front Med (Lausanne). 2021 Jun 16;8:657612. doi: 10.3389/fmed.2021.657612. eCollection 2021. PMID 34222278